CLINICAL TRIAL: NCT06471478
Title: A Retrospective Study Using the Combination of IVIG, Dexamethasone and a Megadose of PBSCs Transfusion for Decreasing DSAs During Haplo-HSCT
Brief Title: The Combination of IVIG, Dexamethasone and a Megadose of PBSCs for Decreasing DSAs
Status: Completed | Type: Observational
Sponsor: Hematology department of the 920th hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KM-05; 202301AY070001-226 (Other Grant/Funding Number: the Joint and Special Project of Kunming medical university)
Record Dates: First submitted 2024-06-13; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Blood Disease
MeSH Terms: conditions — Hematologic Diseases | interventions — Immunoglobulins, Intravenous; Dexamethasone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Combination Product: intravenous immunoglobulin, dexamethasone and a megadose of peripheral-blood stem cell transfusion — patients received intravenous immunoglobulin, dexamethasone and a megadose of peripheral-blood stem cell transfusion for decresing donor specific antibodies.

SUMMARY:
Donor-specific antibodies (DSAs) are essential causes of graft rejection in haploidentical hematopoietic stem cell transplantation (haplo-HSCT). DSAs are unavoidable for some patients who have no alternative donor. Effective interventions to reduce DSAs are still needed, and the cost of the current therapies is relatively high. Investigators wanted to retrospectively analyzed the data of 11 DSA-positive participants who received haplo-HSCT at our center and evaluated the therapeutic efficacy of the combination of intravenous immunoglobulin (IVIG), dexamethasone and megadose of transfused peripheral blood stem cells (PBSCs) for DSA desensitization.

DETAILED DESCRIPTION:
Investigators retrospectively analyzed the data of 11 DSA-positive participants who received haplo-HSCT at our center. All patients received 1 g/kg IVIG on day -1 and 25 mg/m2/d dexamethasone on days -4~-1 before transplantation, and approximately three doses of PBSCs were transfused. On the basis of the conventional transfusion amount of hematopoietic stem cells, additional PBSCs were transfused based on the DSA level of each patient: 3±2×108/kg, 6±2×108/kg and 9±2×108/kg mononuclear cells for participants whose DSAs were weakly positive, positive and strongly positive, respectively.

Blood samples from participants were collected at the following 5 time points: before HSCT and +1 day, +8 day, +15 day and +22 day after transplantation.

The primary endpoint was the incidence of PGF. The secondary endpoints were the incidence of poor graft function, acute and chronic GVHD, relapse, nonrelapse mortality (NRM), overall survival (OS) and disease-free survival (DFS).

ELIGIBILITY:
Inclusion Criteria: DSA positive, receive HSCT in our hospital. -

Exclusion Criteria: Have alternative DSA-negative donor, expended life-span less than 1 month.

-

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received haplo-HSCT and had donor specific antibodies at our hospital were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Graft failure Rate | 2 years
  Number of patients who did not have graft engraftment. Graft failure was defined as the return of recipient hematopoiesis as confirmed by chemerism analysis as <%% donor chimerism at +28 day after HSCT

SECONDARY OUTCOMES:
poor graft function rate | 2 years
  Number of patients who have >95% donor chinerism but blood morphology does not return.
acute graft-versus-host disease rate | 2 years
  the incidence of patients who developed aGVHD
chronic graft-versus-host disease rate | 2 years
  the incidence of patients who developed cGVHD
nonrelapse mortality | 2 years
overall survival | 2 years
disease free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, Professor, Study Director — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Undecided